CLINICAL TRIAL: NCT06255275
Title: Impact of Perceptive, Executive and Emotional Factors on Decision-making in the Context of Pedestrian Crossing in an Industrial Environment Involving Traffic of Autonomous Vehicles (forklifts)
Brief Title: Impact of Perceptive, Executive and Emotional Factors on Decision-making of Pedestrian Face to Autonomous Vehicles.
Acronym: VASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/787
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-04

CONDITIONS: Decision-making

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pedestrian crossing - virtual reality (Experimental)
  Interventions: Other: neurocognitifs tests + pedestrian crossign whith virtual reality

INTERVENTIONS:
Other: neurocognitifs tests + pedestrian crossign whith virtual reality — Neurocognitive tests (attention, executive functions, reaction to difficulty). Assessment of anxiety and impulsivity + pedestrian crossign with virtual reality + post-crossing questionnaire

SUMMARY:
The VASIS project aims to assess the impact of perceptual, executive and emotional factors on decision-making in the context of pedestrian crossing in an industrial environment involving autonomous vehicle traffic (forklift).

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18 to 45
* no objection following submission of a non-objection form indicating that the subject has understood the purpose and procedures of the study and agrees to participate in the study and to comply with the requirements and restrictions inherent in the study

Exclusion Criteria:

* legal incapacity or limited legal capacity
* subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* pregnant or breast-feeding women
* color-blind subject
* history of cardiovascular disease
* current psychiatric or neurological disorders (including self-reported diagnoses of epilepsy)
* known vestibular disorders (prone to frequent dizziness or vertigo)
* headaches or migraines
* deafness
* subjects under the influence of psychotropic substances (alcohol, drugs)
* motor disorders likely to prevent crossing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of the attention of participants on decision-making in the context of pedestrian crossing (virtual reality), particularly on the time required to cross safely, in an industrial environment involving autonomous vehicle traffic. | Day 0
  Quantication of the time required for a pedestrian to cross safely, according to the attention of participants

CONTACTS AND LOCATIONS:
Locations (1):
- Besançon University Hospital, Besançon, France